CLINICAL TRIAL: NCT05527457
Title: Effects of BAY2586116 on Obstructive Sleep Apnoea (OSA) Severity Informed by Upper Airway Physiology and the Role of Route of Breathing
Brief Title: BAY2586116 Nasal Spray and OSA Severity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Flinders University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Professor Danny Eckert, Director, Adelaide Institute for Sleep Health, Flinders University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5468
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and outcomes assessor (sleep scorer) blinded to all 3 study arms. Investigator blinded to 2/3 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo (saline) nasal spray, taken before bedtime. Dosage is taken on one instance for one night only.
  Interventions: Drug: Placebo
- BAY2586116 (oro-nasal breathing night) (Experimental): BAY2586116 nasal spray, taken before bedtime. Dosage is taken on one instance for one night only for the oro-nasal breathing night.
  Interventions: Drug: BAY2586116
- BAY2586116 (nasal breathing only night) (Experimental): BAY2586116 nasal spray, taken before bedtime. Dosage is taken on one instance for one night only for the nasal only breathing night.
  Interventions: Drug: BAY2586116

INTERVENTIONS:
Drug: BAY2586116 — 160 μg BAY2586116 nasal spray application
  Arms: BAY2586116 (nasal breathing only night); BAY2586116 (oro-nasal breathing night)
Drug: Placebo — Placebo (saline) nasal spray application
  Arms: Placebo

SUMMARY:
This investigator-initiated study aims to determine the effects of BAY2586116 (a novel TASK channel blocker nasal spray) on sleep apnoea severity and the potential influence of route of breathing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or older at screening
* Must have completed Part A of the KOALA study (NCT04236440)
* Must be willing to sleep three nights in the sleep lab without OSA therapy (This includes continuous positive airway pressure therapy (CPAP) and/or a mandibular advancement device (MAD))
* Must be willing to refrain from drinking alcohol on the study days.
* Must be willing to limit consumption of tobacco to four cigarettes or one cigar a day and not smoke while at the sleep laboratory. This might be up to 12 hours.
* Must be willing to limit caffeinated beverage intake (coffee, tea, cola, and other soft drinks) to 400 mg / day or less of caffeine and not to be used within 4 hours of bedtime on study days.
* Contraceptive use required by men or women according to the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Any medications or herbal supplements that may interfere or be contraindicated with the study drug as determined by the investigator
* Severely impaired breathing within two days prior to randomization (e.g., acute nasal congestion during upper airway infection).
* known allergies or hypersensitivities to the study drugs (active substances or excipients of the preparations).
* Any other condition which at the discretion of the investigator would make the participant unsuitable for participation in the study and will not allow participation for the full planned study period (e.g., active malignancy or other condition limiting life expectancy to less than 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Individual comparison between physiology changes in Pcrit during KOALA part A (NCT04236440) between BAY2586116 vs. placebo and change in AHI with BAY2586116 vs. placebo (nasal breathing) during current study | Two non-consecutive single night sleep studies (BAY2586116 nasal only breathing night vs. placebo night) conducted approximately 1 week apart
  Individual changes in the critical closing pressure of the upper airway during sleep (Pcrit- measured in cmH2O) in KOALA part A (NCT04236440) will be compared to changes in the apnoea/hypopnoea index (AHI- measured as # of apnoeas and hypopneas per hour of sleep) between BAY2586116 (nasal breathing night) vs. placebo night

SECONDARY OUTCOMES:
Change in OSA severity (BAY2586116 nasal only breathing night vs. placebo night) | Two non-consecutive single night sleep studies (BAY2586116 nasal only breathing night vs. placebo night) conducted approximately 1 week apart
  OSA severity as measured by the AHI (apnoea hypopnea index measured as # events/h sleep) during overnight in-laboratory polysomnography.
Change in OSA severity (BAY2586116 oro-nasal breathing night vs. placebo night) | Two non-consecutive single night sleep studies (BAY2586116 oro-nasal breathing night vs. placebo night) conducted approximately 1 week apart
  OSA severity as measured by the AHI (apnoea hypopnea index measured as # events/h sleep) during overnight in-laboratory polysomnography.
Change in OSA severity (BAY2586116 oro-nasal breathing night vs. BAY2586116 nasal only breathing night) | Two non-consecutive single night sleep studies (BAY2586116 oro-nasal breathing night vs. BAY2586116 nasal only breathing night) conducted approximately 1 week apart
  OSA severity as measured by the AHI (apnoea hypopnea index measured as # events/h sleep) during overnight in-laboratory polysomnography.
Change in nadir overnight hypoxemia (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Nadir overnight oxygen saturation during sleep (%) measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in sleep efficiency (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Percent time spent asleep divided by the recording time from lights out to lights on during overnight in-laboratory polysomnography.
Change in arousal index (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Number of cortical arousals per hour of sleep during overnight in-laboratory polysomnography.
Change in sleep architecture (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Proportion of sleep stages (% total sleep time) during overnight in-laboratory polysomnography.
Change in respiratory control (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Loop gain and the ventilatory response to arousal (% eupnea) during overnight in-laboratory polysomnography.
Change in the respiratory arousal threshold (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Threshold to arousal (% eupnea) during overnight in-laboratory polysomnography.
Change in airway collapsibility (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Vpassive (% eupnea) during overnight in-laboratory polysomnography.
Placebo OSA endotypes (outcomes 8-11) and whether they are associated with changes in OSA severity (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Exploratory analysis to determine if OSA endotypes (outcomes 8-11) are associated with changes in OSA severity (BAY2586116 nights vs. placebo night)
Change in hypoxic burden (BAY2586116 nights vs. placebo night) | Three non-consecutive single night sleep studies (BAY2586116 nasal only breathing night, BAY2586116 oro-nasal breathing night and placebo night) conducted approximately 1 week apart
  Hypoxic burden during sleep (%min/h) measured via pulse oximetry during overnight in-laboratory polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Danny J. Eckert, PhD, Principal Investigator — Flinders University
Locations (1):
- Flinders University, Bedford Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be included in the study publication.
Supporting Information: Study Protocol
Time Frame: Upon publication
Access Criteria: Available in the publication.

REFERENCES:
- [Background] Gaisl T, Turnbull CD, Weimann G, Unger S, Finger R, Xing C, Cistulli PA, West S, Chiang AKI, Eckert DJ, Stradling JR, Kohler M. BAY 2253651 for the treatment of obstructive sleep apnoea: a multicentre, double-blind, randomised controlled trial (SANDMAN). Eur Respir J. 2021 Nov 18;58(5):2101937. doi: 10.1183/13993003.01937-2021. Print 2021 Nov. PMID 34531274
- See also: Clinical trial registry for main KOALA study protocol (Parts A-C) — https://clinicaltrials.gov/ct2/show/NCT04236440